CLINICAL TRIAL: NCT03012672
Title: Impact of Treatment Intensity on Survival, Quality of Life, and Resource Utilization in Medically Less Fit Adults With Acute Myeloid Leukemia and Analogous Myeloid Neoplasms: A Randomized Pilot Study
Brief Title: Higher or Lower Dose Cladribine, Cytarabine, and Mitoxantrone in Treating Medically Less Fit Patients With Newly Diagnosed Acute Myeloid Leukemia or Myeloid Neoplasm
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Anna Halpern, Assistant Professor, Division of Hematology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9759; NCI-2016-02051 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9759 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); RG9217016 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2017-01-03; First posted 2017-01-06 (Estimated); Results first posted 2021-11-01 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Acute Leukemia of Ambiguous Lineage; Acute Myeloid Leukemia; Myeloid Neoplasm
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Leukemia, Myeloid, Acute | interventions — Cladribine; Cytarabine; Granulocyte Colony-Stimulating Factor; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (higher-dose) (Experimental): INDUCTION: Patients receive G-CSF SC on days 0-5, higher dose cladribine IV over 2 hours on days 1-5, higher dose cytarabine IV over 2 hours on days 1-5, and higher dose mitoxantrone IV over 60 minutes on days 1-3. Treatment repeats every 6 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients who achieve CR/CRi with up to 2 courses of Induction receive G-CSF, cladribine, and cytarabine as in Induction. Courses repeat every 6 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cladribine; Drug: Cytarabine; Biological: Granulocyte Colony-Stimulating Factor; Drug: Mitoxantrone Hydrochloride; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (lower-dose) (Experimental): INDUCTION: Patients receive G-CSF SC on days 0-5, lower dose cladribine IV over 2 hours on days 1-5, lower dose cytarabine IV over 1 hour on days 1-5, and lower dose mitoxantrone IV over 60 minutes on days 1-3. Treatment repeats every 6 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients who achieve CR/CRi with up to 6 courses of Induction receive G-CSF, cladribine, and cytarabine as in Induction. Courses repeat every 6 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cladribine; Drug: Cytarabine; Biological: Granulocyte Colony-Stimulating Factor; Drug: Mitoxantrone Hydrochloride; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Cladribine — Given IV
  Other Names: 2-CdA; 2CDA; CdA; Cladribina; Leustat; Leustatin; Leustatine; RWJ-26251
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosar-U; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Biological: Granulocyte Colony-Stimulating Factor — Given SC
  Other Names: Colony Stimulating Factor 3; Colony-Stimulating Factor (Granulocyte); Colony-Stimulating Factor 3; CSF3; G CSF; G-CSF; Granulocyte Colony Stimulating Factor; Pluripoietin
Drug: Mitoxantrone Hydrochloride — Given IV
  Other Names: CL 232315; DHAD; DHAQ; Dihydroxyanthracenedione Dihydrochloride; Mitoxantrone Dihydrochloride; Mitoxantroni Hydrochloridum; Mitozantrone Hydrochloride; Mitroxone; Neotalem; Novantrone; Onkotrone; Pralifan
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized pilot trial studies how well higher or lower dose cladribine, cytarabine, and mitoxantrone work in treating medically less fit patients with newly diagnosed acute myeloid leukemia or myeloid neoplasm. Drugs used in chemotherapy, such as cladribine, cytarabine, and mitoxantrone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether giving cladribine, cytarabine, and mitoxantrone at higher or lower dose may work better in treating patients with newly diagnosed acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the feasibility of randomizing medically less fit adults with newly diagnosed acute myeloid leukemia (AML) or analogous myeloid neoplasms to either intensive or non-intensive induction and post remission chemotherapy.

EXPLORATORY OBJECTIVES:

I. To evaluate the attitude of patients and physicians toward randomization and explore reasons for treatment preference.

II. To evaluate whether the ability to assess fitness for intensive chemotherapy can be improved by an augmented treatment-related mortality (TRM) score that includes additional (co-morbidity) factors, and to compare the ability of physicians and the prediction algorithm(s) to assess the likelihood of early death.

III. To compare, within the limits of a pilot study, response, duration of response, and survival between patients receiving intensive and those receiving non-intensive chemotherapy.

IV. To describe the impact of treatment intensity on quality of life of patients undergoing chemotherapy for newly diagnosed AML.

V. To describe the impact of treatment intensity on medical resource utilization and care cost of patients undergoing chemotherapy for newly diagnosed AML.

OUTLINE: Patients agreeable to randomization are randomized to 1 of 2 treatment arms. Patients not agreeable to randomization receive treatment based on their preference.

ARM I (HIGHER-DOSE):

INDUCTION: Patients receive granulocyte colony-stimulating factor (G-CSF) subcutaneously (SC) on days 0-5, higher dose cladribine intravenously (IV) over 2 hours on days 1-5, higher dose cytarabine IV over 2 hours on days 1-5, and higher dose mitoxantrone IV over 60 minutes on days 1-3. Treatment repeats every 6 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION: Patients who achieve complete response (CR)/CR with incomplete count recovery (CRi) with up to 2 courses of Induction receive G-CSF, cladribine, and cytarabine as in Induction. Courses repeat every 6 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.

ARM II (LOWER-DOSE):

INDUCTION: Patients receive G-CSF SC on days 0-5, lower dose cladribine IV over 2 hours on days 1-5, lower dose cytarabine IV over 1 hour on days 1-5, and lower dose mitoxantrone IV over 60 minutes on days 1-3. Treatment repeats every 6 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION: Patients who achieve complete response (CR)/CR with incomplete count recovery (CRi) with up to 6 courses of Induction receive G-CSF, cladribine, and cytarabine as in Induction. Courses repeat every 6 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of untreated "high-grade" myeloid neoplasm (>= 10% myeloid blasts by morphology in bone marrow and/or peripheral blood) or AML other than acute promyelocytic leukemia (APL) with t(15;17)(q22;q12) or variants according to the 2016 World Health Organization (WHO) classification; patients with acute leukemias of ambiguous lineage are eligible; outside diagnostic material is acceptable as long as peripheral blood and/or bone marrow slides are reviewed at the study institution and cytogenetic/molecular information is available
* Treatment-related mortality (TRM) score >= 13.1 as calculated with simplified model
* The use of hydroxyurea before enrollment is permitted; hydroxyurea should be discontinued prior to start of study treatment. Patients with symptoms/signs of leukostasis, white blood cell (WBC) > 100,000/uL, or acute symptoms felt related to their high-grade myeloid neoplasm can be treated with leukapheresis or may receive up to 1 dose of cytarabine (up to 500 mg/m^2) anytime prior to study day 1
* Patients may have received treatment (e.g. azacitidine/decitabine, lenalidomide, growth factors) for antecedent low-grade myeloid neoplasm
* Left ventricular ejection fraction (LVEF) >= 45%, assessed within 3 months prior to registration, e.g. by multigated acquisition (MUGA) scan or echocardiography, or other appropriate diagnostic modality
* Women of childbearing potential and men must agree to use adequate contraception beginning at the signing of the consent until at least 4 weeks after the last dose of study drug
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Myeloid blast crisis of chronic myeloid leukemia (CML), unless patient is not considered candidate for tyrosine kinase inhibitor treatment
* Concomitant illness associated with a likely survival of < 1 year
* Active systemic fungal, bacterial, viral, or other infection, unless disease is under treatment with anti-microbials and/or controlled or stable; patients with fever thought to be likely secondary to leukemia are eligible; known hypersensitivity to any study drug
* Known hypersensitivity to any study drug used in this trial
* Pregnancy or lactation
* Concurrent treatment with any other anti-leukemia agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-12-30 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2021-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Halpern, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Higher-dose) | Arm II (Lower-dose)
Started | 20 | 30
Completed | 20 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ARM I (HIGHER-DOSE): ARM I (HIGHER-DOSE):
  INDUCTION: Patients receive granulocyte colony-stimulating factor (G-CSF) subcutaneously (SC) on days 0-5, higher dose cladribine intravenously (IV) over 2 hours on days 1-5, higher dose cytarabine IV over 2 hours on days 1-5, and higher dose mitoxantrone IV over 60 minutes on days 1-3. Treatment repeats every 6 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients who achieve complete response (CR)/CR with incomplete count recovery (CRi) with up to 2 courses of Induction receive G-CSF, cladribine, and cytarabine as in Induction. Courses repeat every 6 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.
- ARM II (LOWER-DOSE): ARM II (LOWER-DOSE):
  INDUCTION: Patients receive G-CSF SC on days 0-5, lower dose cladribine IV over 2 hours on days 1-5, lower dose cytarabine IV over 1 hour on days 1-5, and lower dose mitoxantrone IV over 60 minutes on days 1-3. Treatment repeats every 6 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients who achieve complete response (CR)/CR with incomplete count recovery (CRi) with up to 6 courses of Induction receive G-CSF, cladribine, and cytarabine as in Induction. Courses repeat every 6 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | ARM I (HIGHER-DOSE) | ARM II (LOWER-DOSE) | Total
Number analyzed (Participants) | 20 | 30 | 50
Age, Continuous [Median (Full Range); unit: years] | 71.5 [42 to 82] | 72 [44 to 89] | 72 [42 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 12 | 21 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 2 | 2
  White | 19 | 25 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Secondary Disease [Count of Participants; unit: Participants]
  De Novo | 10 | 15 | 25
  Secondary | 10 | 15 | 25
ELN Risk Category [Count of Participants; unit: Participants]
  Favorable | 1 | 3 | 4
  Intermediate | 5 | 6 | 11
  Adverse | 9 | 17 | 26
  No Classifiable | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Feasibility Defined as Proportion of Patients Willing to be Randomized to Either Intensive or Non-intensive Induction and Post Remission Chemotherapy
Description: Randomizing patients to either intensive or non-intensive induction and post remission chemotherapy will be considered feasible if the true proportion of patients willing to be randomized is 60% or higher.
Time Frame: At end of enrollment
Measure: Count of Participants; unit: Participants
Groups:
- All Patients Enrolled: Total number of patients enrolled
Arm/Group | All Patients Enrolled
Number analyzed (Participants) | 50
Participants
  Patients/physician pairs agreed to be randomized | 3
  Patients/physician pairs not agreed to be randomized | 47

2. Other Pre Specified Outcome: Event-free Survival
Description: Will be determined by peripheral blood count and bone marrow evaluation and categorized according to criteria recommended by International Working Groups.
Time Frame: Up to 5 years
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Medical Complications
Description: Information on medical complications (e.g. need for intensive care unit (ICU) level care, length of ICU stay, neutropenic fever, documented infections, bleeding, reasons for hospitalization) will be collected from the medical records from the University of Washington Medical Center (UWMC) and Seattle Cancer Care Alliance (SCCA).
Time Frame: Up to 5 years
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Medical Resource Utilization
Description: Information on use of medical resources (e.g. platelet transfusions; days of IV antimicrobial therapy, total hospital length of stay) will be collected from the medical records from the University of Washington Medical Center (UWMC) and Seattle Cancer Care Alliance (SCCA).
Time Frame: Up to 5 years
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Overall Survival
Description: Will be assessed for all patients. Will be determined by peripheral blood count and bone marrow evaluation and categorized according to criteria recommended by International Working Groups.
Time Frame: Up to 5 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Quality of Life as Measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30
Description: Will be measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30. Exploratory, descriptive, and observational methods will be used.
Time Frame: Up to 12 months
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Relapse-free Survival
Description: as for outcome 2
Time Frame: Up to 5 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Response
Description: The differences in anti-leukemic efficacy between patients treated with lower-intensity chemotherapy and those treated with higher-intensity chemotherapy will be estimated. Exploratory, descriptive, and observational methods will be used.
Time Frame: Up to 5 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Fitness for Intensive Chemotherapy as Measured by a Treatment-related Mortality (TRM) Score That Includes Additional Co-morbidity Factors
Description: The ability of physicians and the prediction algorithm(s) to assess the likelihood of early death will be compared.
Time Frame: Up to 12 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Duration of Response
Description: Will be evaluated.
Time Frame: Up to 5 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Care Costs
Description: The costs associated with inpatient and outpatient management will be calculated using electronic billing information from the University of Washington Medical Center (UWMC) and Seattle Cancer Care Alliance (SCCA). Costs will be converted from charges using departmental cost-to-charge ratios. Descriptive information identifying major cost drivers and total/subset costs per phase of treatment will be reported.
Time Frame: Up to 5 years
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Attitude of Patients Toward Randomization
Description: Will be determined by a patient preference survey. Exploratory, descriptive, and observational methods will be used.
Time Frame: Up to 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: AEs were collected for the duration that each patient remained on protocol. If a subject decided to terminate the study early AEs continued to be collected for up to 4 weeks after the treatment was given or until they started a new anti-leukemia therapy, whichever occurred first.
Description: Only grade ≥3 adverse events other than hematologic toxicities were recorded, graded, and reported as appropriate.
Groups:
- ARM I (HIGHER-DOSE):: ARM I (HIGHER-DOSE):
  INDUCTION: Patients receive granulocyte colony-stimulating factor (G-CSF) subcutaneously (SC) on days 0-5, higher dose cladribine intravenously (IV) over 2 hours on days 1-5, higher dose cytarabine IV over 2 hours on days 1-5, and higher dose mitoxantrone IV over 60 minutes on days 1-3. Treatment repeats every 6 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients who achieve complete response (CR)/CR with incomplete count recovery (CRi) with up to 2 courses of Induction receive G-CSF, cladribine, and cytarabine as in Induction. Courses repeat every 6 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.
- ARM II (LOWER-DOSE):: ARM II (LOWER-DOSE):
  INDUCTION: Patients receive G-CSF SC on days 0-5, lower dose cladribine IV over 2 hours on days 1-5, lower dose cytarabine IV over 1 hour on days 1-5, and lower dose mitoxantrone IV over 60 minutes on days 1-3. Treatment repeats every 6 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients who achieve complete response (CR)/CR with incomplete count recovery (CRi) with up to 6 courses of Induction receive G-CSF, cladribine, and cytarabine as in Induction. Courses repeat every 6 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | ARM I (HIGHER-DOSE): | ARM II (LOWER-DOSE):
All-Cause Mortality (participants affected / at risk) | 16/20 | 25/30
Serious Adverse Events (participants affected / at risk) | 9/20 | 14/30
Other Adverse Events (participants affected / at risk) | 16/20 | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM I (HIGHER-DOSE): (N=20) | ARM II (LOWER-DOSE): (N=30)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
Intracranial Hemorrhage (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 2 (2)
Febrile Neutropenia (Blood and lymphatic system disorders) | 6 (8) | 7 (13)
Lung Infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Right Ventricular Dysfunction (Cardiac disorders) | 1 (1) | 0 (0) — Type II NSTEMI
Delirium (Psychiatric disorders) | 2 (2) | 0 (0)
Vascular Access Complication (Vascular disorders) | 1 (1) | 0 (0) — Non-occlusive R axillary DVT and superficial thrombophlebitis
Generalized Edema (General disorders) | 1 (1) | 0 (0) — Anasarca
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Colonic Pseudo-Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM I (HIGHER-DOSE): (N=20) | ARM II (LOWER-DOSE): (N=30)
Acute Kidney Injury (Renal and urinary disorders) | 1 (2) | 2 (2)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 2 (3) | 1 (1)
Bacteremia (Infections and infestations) | 5 (5) | 4 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Blood Clot, Right Ear (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Edema Limbs, Volume Overload (Cardiac disorders) | 2 (2) | 2 (2)
Epistaxis (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Febrile Neutropenia (Blood and lymphatic system disorders) | 9 (10) | 15 (21)
AST/ALT Elevation (Investigations) | 0 (0) | 1 (1)
Blood Bilirubin Increased (Investigations) | 2 (2) | 1 (1)
Bronchopulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cardiac Troponin I Increased (Cardiac disorders) | 3 (4) | 2 (2)
Catheter Related Infection (Infections and infestations) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 2 (2) | 1 (1)
Ejection Fraction Decreased (Investigations) | 0 (0) | 1 (1)
Generalized Edema (General disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypertension (Cardiac disorders) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 9 (9)
Lung Infection (Infections and infestations) | 1 (1) | 4 (5)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Optic Nerve Disorder (Eye disorders) | 1 (1) | 0 (0)
Paroxysmal Atrial Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 8 (8)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 4 (4) | 4 (4)
Soft Tissue Infection (Infections and infestations) | 2 (2) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 2 (3) | 4 (4)
Mucositis (Infections and infestations) | 0 (0) | 1 (1)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Restrictive Cardiomyopathy (Cardiac disorders) | 0 (0) | 2 (2)
Tumor Lysis Syndrome (Blood and lymphatic system disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-20): https://cdn.clinicaltrials.gov/large-docs/72/NCT03012672/Prot_SAP_000.pdf